CLINICAL TRIAL: NCT02511977
Title: Evaluation Clinical and Radiographic Images in Dental Implants Rehabilitated With Overdentures
Status: Completed | Type: Observational
Sponsor: Universidade Metropolitana de Santos (Other)
Responsible Party: Principal Investigator, CAIO VINICIUS GONÇALVES ROMAN TORRES, Principal investigator, Universidade Metropolitana de Santos
Other Study IDs: SANTOSMU02
Record Dates: First submitted 2015-06-05; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Failure of Dental Implant Due to Lack of Attached Gingiva; Failure of Dental Prosthesis Causing Loss of Dental Implant
Keywords: Dental Prosthesis; Implant-Supported

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- overdenture with annual maintenance: Rehabilitation should be: overdenture with at least 2 implants placed in the mandible and 3 implants in the maxilla per person. They were divided into two groups: Group I: Annual maintenance for the past seven years
  Interventions: Other: peri-implant examination
- overdenture whitout annual maintenance: Group II: individuals who have not returned for the last seven years. Individuals who said they went to the dentist at least once a year, for whatever treatment, were included in the maintenance group. Individuals who denied any visit to the dentist in the last seven years were included in the no maintenance group.
  Interventions: Other: peri-implant examination

INTERVENTIONS:
Other: peri-implant examination — The prostheses were removed and all implants were evaluated: probing depth, plaque index and bleeding index.

SUMMARY:
The control of biofilm around implants is critical to the success of the implant rehabilitation of edentulous jaw with overdentures, and it is the dentist's duty to inform and guide patients, and keep their maintenance in order to prevent pathological processes that can lead to the implanted component loss.The aim of the present retrospective longitudinal study was to evaluate through clinical periodontal parameters and radiographic images in dental implants rehabilitated with overdentures installed seven years ago. individuals who underwent the installation of dental implants for making full implant-supported upper and lower mucus dentures in the Department of Implant Dentistry, Faculty of Dentistry, University of Santo Amaro, São Paulo, Brazil, in 2007. The periodontal parameters such as probing depth, plaque index, bleeding index and mobility as well as radiographic examination, are key to determine the correct diagnosis in dental implants. The control of biofilm around the implants seems to be a decisive factor for maintaining tissue health. We believe that the maintenance appointments are fundamental, but more studies should be conducted to elucidate microbial and immunological factors in implants placed and due for some time.

DETAILED DESCRIPTION:
The control of biofilm around implants is critical to the success of the implant rehabilitation of edentulous jaw with overdentures, and it is the dentist's duty to inform and guide patients, and keep their maintenance in order to prevent pathological processes that can lead to the implanted component loss.The aim of the present retrospective longitudinal study was to evaluate through clinical periodontal parameters and radiographic images in dental implants rehabilitated with overdentures installed seven years ago. individuals who underwent the installation of dental implants for making full implant-supported upper and lower mucus dentures in the Department of Implant Dentistry, Faculty of Dentistry, University of Santo Amaro, São Paulo, Brazil, in 2007. The periodontal parameters such as probing depth, plaque index, bleeding index and mobility as well as radiographic examination, are key to determine the correct diagnosis in dental implants. The control of biofilm around the implants seems to be a decisive factor for maintaining tissue health.

ELIGIBILITY:
Inclusion Criteria:

* Rehabilitation should be:prothesis type overdenture, with at least 2 implants placed in the mandible and 3 implants in the maxilla per person
* individuals who have annual maintenance for the past seven years,
* individuals who have not returned for the last seven years,
* Individuals who said they went to the dentist at least once a year, for whatever treatment, were included in the maintenance group,
* Individuals who denied any visit to the dentist in the last seven years were included in the no maintenance group.

Exclusion Criteria:

* smokers,
* as those who, for any reason, should make systemic medication suspension for clinical evaluation,
* individuals in need of antibiotic prophylaxis for carrying out the clinical examinations,
* Patients with less than seven annual maintenance consultations in the last seven years

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Initially, 80 individuals who underwent the installation of dental implants for making overdentures in the Department of Implant Dentistry, Faculty of Dentistry, University of Santo Amaro, São Paulo, Brazil, in 2007,were evaluated.According to the inclusion and exclusion criteria, the final sample had 64 individuals of both genders, between 40 and 75 years old
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
probing depth in implants | 7 years
  individuals who underwent the installation of dental implants for making full upper and lower overdentures in 2007

SECONDARY OUTCOMES:
gingival index (GI) | 7 years
  individuals who underwent the installation of dental implants for making full upper and lower overdentures in 2007
plaque index (PI) | 7 years
  individuals who underwent the installation of dental implants for making full upper and lower overdentures in 2007

CONTACTS AND LOCATIONS:
Overall Officials: Caio VG Roman-Torres, PhD, Principal Investigator — University of South Australia
Locations (1):
- University of Santo Amaro - UNISA/SP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Meijer HJ, Raghoebar GM, de Waal YC, Vissink A. Incidence of peri-implant mucositis and peri-implantitis in edentulous patients with an implant-retained mandibular overdenture during a 10-year follow-up period. J Clin Periodontol. 2014 Dec;41(12):1178-83. doi: 10.1111/jcpe.12311. Epub 2014 Nov 1. PMID 25229397
- [Result] Parmar S, Karir N, Walmsley D, Patel U. Long and short term management of implant-supported mandibular overdentures. Dent Update. 2013 Dec;40(10):830-2, 834-5. doi: 10.12968/denu.2013.40.10.830. PMID 24597027
- [Result] Troeltzsch M, Troeltzsch V, Brodine AH, Frankenberger R, Messlinger K, Troeltzsch M. Clinical performance and peri-implant parameters of 132 implants supporting locator-retained overdentures: a case series of 33 patients. Int J Oral Maxillofac Implants. 2013 Jul-Aug;28(4):1132-9. doi: 10.11607/jomi.3009. PMID 23869372
- [Result] Akca K, Cehreli MC, Uysal S. Marginal bone loss and prosthetic maintenance of bar-retained implant-supported overdentures: a prospective study. Int J Oral Maxillofac Implants. 2010 Jan-Feb;25(1):137-45. PMID 20209196
- [Result] Cehreli MC, Uysal S, Akca K. Marginal bone level changes and prosthetic maintenance of mandibular overdentures supported by 2 implants: a 5-year randomized clinical trial. Clin Implant Dent Relat Res. 2010 Jun 1;12(2):114-21. doi: 10.1111/j.1708-8208.2008.00143.x. Epub 2009 Feb 13. PMID 19220845